CLINICAL TRIAL: NCT05450341
Title: Efficacy of Low-frequency Repetitive Transcranial Magnetic Stimulation on Rehabilitation of Aphasia
Brief Title: Efficacy of Low-frequency rTMS in Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Talat Bulut, Assist. Prof. Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Aphasia
Keywords: Repetitive transcranial magnetic stimulation; Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: The two groups receive one of the two treatments: right frontal versus right temporal stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcomes assessor (speech and language therapist conducting the assessment tests and the eyetracking experiment) will be blind as to which experiment group the participant belongs to. The investigator / clinician providing rTMS will not be blind to the experimental condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right frontal 1 Hz rTMS (Experimental): Low-frequency (1 Hz) inhibitory rTMS will be administered to right inferior frontal gyrus with the following parameters:
  Frequency: 1 Hz Stimulation site: Right IFG (as determined using EEG 10-20 system) Intensity: 100% of motor threshold Dosage: 20 minutes per day Duration: 10 days over 2 weeks (no stimulation during weekends)
  Interventions: Device: rTMS over right frontal target
- Right temporal 1 Hz rTMS (Active Comparator): Low-frequency (1 Hz) inhibitory rTMS will be administered to right posterior superior temporal gyrus with the following parameters:
  Frequency: 1 Hz Stimulation site: Right posterior superior temporal gyrus (as determined using EEG 10-20 system) Intensity: 100% of motor threshold Dosage: 20 minutes per day Duration: 10 days over 2 weeks (no stimulation during weekends)
  Interventions: Device: rTMS over right temporal target

INTERVENTIONS:
Device: rTMS over right frontal target — Low frequency (1 Hz) rTMS over right inferior frontal gyrus
  Arms: Right frontal 1 Hz rTMS
Device: rTMS over right temporal target — Low frequency (1 Hz) rTMS over right posterior superior temporal gyrus
  Arms: Right temporal 1 Hz rTMS

SUMMARY:
In a randomized controlled trial, efficacy of low-frequency, inhibitory rTMS will be examined in rehabilitation of acquired aphasia. Two cortical sites will be targeted: Right-hemispheric homologues of Broca's and Wernicke's areas.

In addition to cognitive screening prior to onset of rTMS, language assessments will be conducted before, during and after the intervention. An eyetracking-while-listening experiment will also be conducted before and after the intervention to investigate morphosyntactic processing.

DETAILED DESCRIPTION:
Efficacy of low-frequency (1hz), inhibitory rTMS will be examined in rehabilitation of acquired aphasia. Two cortical sites will be targeted: Right-hemispheric homologues of Broca's and Wernicke's areas. In other words, right frontal and right temporal sites will be targeted.

In addition to cognitive screening prior to onset of rTMS, language assessments will be conducted before, during and after the intervention. The language assessment will be conducted using the Turkish Aphasia Language Assessment Test (ADD) and sets of pictures used to assess naming performance. ADD will be carried out before and after the intervention. Six picture sets will be used, one at baseline, four on different days during the intervention, and the last one immediately after the last day of the intervention. Cognitive screening will be conducted at baseline using the digit span test and Raven's colored progressive matrices. In addition, a pre- and post-treatment eyetracking-while-listening experiment will be conducted to investigate morphosyntactic processing in Turkish and to examine whether the two brain stimulation interventions differentially affect online (dynamic, time-dependent) measures of morphosyntactic processing. The eyetracking paradigm will request the participants to listen to Turkish sentences varying in morphosyntactic complexity (canonical versus noncanonical sentences) and to look at the picture (out of two pictures presented on the screen) corresponding to the sentence they are listening to.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness,
* Normal or corrected-to-normal vision and hearing,
* Aphasia following cerebrovascular accident,
* Cerebrovascular accident at least 6 months prior to enrolment in the study,
* Satisfying current TMS safety guidelines (Rossi et al. 2009, 2021), which are:
* No previous history of epilepsy,
* No implant (e.g., cochlear implant) or stimulator (e.g., deep brain stimulation) in the head which may interact with the magnetic field,
* No use of central nervous system active drugs that lower seizure threshold (as listed in the aforementioned guidelines)

Exclusion Criteria:

* Left-handedness, ambidexterity,
* Impaired and uncorrected vision or hearing,
* No aphasia symptoms following cerebrovascular accident,
* Time since cerebrovascular accident less than 6 months,
* Violating current TMS safety guidelines (Rossi et al. 2009, 2021). In other words:
* Having a previous history of epilepsy,
* Having an implant (e.g., cochlear implant) or stimulator (e.g., deep brain stimulation) in the head which may interact with the magnetic field,
* Taking central nervous system active drugs that lower seizure threshold (as listed in the aforementioned guidelines)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Turkish Aphasia Language Assessment Test Scores Time 1 (pre-treatment) | Immediately before the intervention (Day 0)
  Baseline scores obtained from the Turkish Aphasia Language Assessment Test (ADD) Minimum score: 0 points Maximum score: 292 points Higher scores indicate a better outcome
Turkish Aphasia Language Assessment Test Scores Time 2 (during treatment) | At the end of the first week of intervention (Day 5)
  Scores obtained from the Turkish Aphasia Language Assessment Test (ADD) at the end of the first week of treatment Minimum score: 0 points Maximum score: 292 points Higher scores indicate a better outcome
Turkish Aphasia Language Assessment Test Scores Time 3 (post-treatment short-term) | Immediately after the intervention (Day 10)
  Post-treatment scores obtained from the Turkish Aphasia Language Assessment Test (ADD) at the end of the treatment Minimum score: 0 points Maximum score: 292 points Higher scores indicate a better outcome
Turkish Aphasia Language Assessment Test Scores Time 4 (post-treatment medium-term) | 1 month after the intervention
  Post-treatment scores obtained from the Turkish Aphasia Language Assessment Test (ADD) one month after the end of the treatment Minimum score: 0 points Maximum score: 292 points Higher scores indicate a better outcome
Turkish Aphasia Language Assessment Test Scores Time 5 (post-treatment long-term) | 6 months after the intervention
  Post-treatment scores obtained from the Turkish Aphasia Language Assessment Test (ADD) six months after the end of the treatment Minimum score: 0 points Maximum score: 292 points Higher scores indicate a better outcome
Picture Naming Scores Time 1 (pre-treatment) | Immediately before the intervention (Day 0)
  Picture naming performance (number of accurately named pictures & naming latency for correctly named pictures) There are 20 pictures in total, of which half are objects and half actions. Minimum score: 0 points Maximum score: 20 points Higher scores indicate a better outcome
Picture Naming Scores Time 2 (during treatment) | At the end of the first week of intervention (Day 5)
  Picture naming performance (number of accurately named pictures & naming latency for correctly named pictures) There are 20 pictures in total, of which half are objects and half actions. Minimum score: 0 points Maximum score: 20 points Higher scores indicate a better outcome
Picture Naming Scores Time 3 (post-treatment short-term) | Immediately after the intervention (Day 10)
  Picture naming performance (number of accurately named pictures & naming latency for correctly named pictures) There are 20 pictures in total, of which half are objects and half actions. Minimum score: 0 points Maximum score: 20 points Higher scores indicate a better outcome
Picture Naming Scores Time 4 (post-treatment medium-term) | 1 month after the intervention
  Picture naming performance (number of accurately named pictures & naming latency for correctly named pictures) There are 20 pictures in total, of which half are objects and half actions. Minimum score: 0 points Maximum score: 20 points Higher scores indicate a better outcome
Picture Naming Scores Time 5 (post-treatment long-term) | 6 months after the intervention
  Picture naming performance (number of accurately named pictures & naming latency for correctly named pictures) There are 20 pictures in total, of which half are objects and half actions. Minimum score: 0 points Maximum score: 20 points Higher scores indicate a better outcome
Eye movements Time 1 (pre-treatment) | Immediately before the intervention (Day 0)
  An eyetracking-while-listening paradigm will be used to determine proportions of dwell time on the correct picture (out of two alternatives) corresponding to auditorily presented Turkish sentences varying in morphosyntactic complexity.
Eye movements Time 2 (post-treatment) | Immediately after the intervention (Day 10)
  An eyetracking-while-listening paradigm will be used to determine proportions of dwell time on the correct picture (out of two alternatives) corresponding to auditorily presented Turkish sentences varying in morphosyntactic complexity.

CONTACTS AND LOCATIONS:
Overall Officials: Talat Bulut, Ph.D., Principal Investigator — Medipol University
Locations (1):
- İstanbul Medipol University, Speech, Language and Swallowing Therapy and Research Center (MEDKOM), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants' anonymized data will be shared with the scientific community as part of open science practices. IPD refer to the data collected from the participants (language and cognitive test scores; i.e., ADD and naming performance, number/percentage of correct answers, raw and scaled scores, short-term memory scores (digit span), nonverbal intelligence scores (Raven's colored progressive matrices). IPD also include eye movements data obtained in the eyetracking experiment; i.e., proportions of dwell time on the target picture.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication of the results in a peer-reviewed journal. The data will be shared permanently.
Access Criteria: No access criteria required; a permanent link to the dataset will be made available so that the public can access the data (e.g., using https://osf.io/ or Mendeley Data)

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT05450341/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT05450341/ICF_001.pdf